CLINICAL TRIAL: NCT06419426
Title: Studio Prospettico Sulle Batteriemie Febbrili Nei Pazienti Oncoematologici Pediatrici
Brief Title: Prospective Study on Febrile Batteries in Pediatric Oncohaematological Patients (SuBiTo)
Acronym: SuBiTo
Status: Active, not recruiting | Type: Observational
Sponsor: Associazione Italiana Ematologia Oncologia Pediatrica (Other)
Responsible Party: Sponsor
Other Study IDs: SuBiTO
Record Dates: First submitted 2021-03-08; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Battery incidence — Incidence of batteries from negative Gram germs; Incidence of batteries from gram positive germs; Incidence of fungemie; Incidence of septic shock; Incidence of batteries from colonising germs; Incidence of resistance to the main classes of antibiotics

SUMMARY:
The aim of this study is to define prospectively the incidence of multi-resistant germ batteries in paediatric oncoematological patients, to assess associated mortality, antibiotic resistance profile and the type of implemented therapy.

DETAILED DESCRIPTION:
Bacterial infections are the most frequent cause of infectious morbidity and mortality in the patient undergoing chemotherapy or hemopoietic stem cell transplantation (TCSE). The main predisposing factor is the impairment of innate immunity as a result of the alteration of mucous barriers (mucositis/enteritis from chemotherapy or radiotherapy), skin (CVC) and neutropenia (non-specific haematological toxicity due to chemotherapy or radiotherapy on bones with hemopoietic marrow). The most frequent form of infection is represented by fever whose cause remains indeterminate in 60-80% of cases. In about 10-15% of cases fever is accompanied by the positivization of hemoculture and is configured as a microbiologically determined infection (IMD). In the remaining cases, infectious episodes may be clinically documented such as pneumonia or bronchitis confirmed for radiological examination or CT scans, without the identification of the causative agent; these are defined as clinically determined infections (ICDs).

The knowledge, through hemoculture, of the germs responsible for febrile batteries over a given period of time, allows the definition of the predominant typology of germs responsible for systemic infection. On this basis, it is used to define the empirical antibiotic treatment that is given to the patient within a few hours of the onset of fever. Empirical antibiotic therapy must be effective with regard to the germs most represented in the department or in the area in question. Once the result of hemoculture has been received, usually within 48-72 hours, empirical antibiotic therapy can be maintained or modified in relation to the type of isolated germ and its susceptibility to antibiotics included in the empirical scheme. In fact, there is ample evidence that ready-to-treat with broad-spectrum antibiotics reduces mortality from bacterial infection in the immunocompromised patient, so this procedure is now a recommended approach by the guidelines. In addition to the knowledge of prevalent bacterial epidemiology for a certain type of immunocompromised patients in a given geographical area, a second tool capable of allowing appropriate empirical antibiotic therapy is the choice of therapy based on the presence or not of asymptomatic bacterial colonization of the patient. In fact, it is estimated that in 20-30% of cases the colonizing germ can become the cause of a batteriemia, facilitated by favoring factors such as the rupture of skin-mucous reefs or the appearance of neutropenia. The need to start empirical antibiotic therapy with effective molecules against causal germ (appropriate empirical therapy) has been shown to reduce bacterial infectious mortality at a time when antibiotic resistance is gradually increasing. It has been shown that inappropriate empirical antibiotic therapy, based on antibiotics to which the germ is not sensitive, is associated with increased infectious mortality from sepsis and septic shock. Among the adjuvant therapies used in immunosuppressed patients, in addition to antibiotic therapy, especially in patients with septic shock, there is the administration of opsonizing immunoglobulins and able to activate the complement such as, for example, immunoglobulins enriched in IgM. This practice is generally more established in immunocompetent patients while there are no prospective data in immunocompromised patients.

Primary objective Incidence of febrile batteries from antibiotic-resistant gram negative germs (MDR)

Secondary objectives Incidence of batteries from negative Gram germs; Incidence of batteries from gram positive germs; Incidence of fungemie; Incidence of septic shock; Incidence of batteries from colonising germs; Incidence of resistance to the main classes of antibiotics used empirically: cephalosporins of 3 and 4 generation (ceftazidime, cefipime), semisitical penicillins (piperacillin/tazobactam), carbapenemas (meropenem, imipenem), aminoglycosides (aminoglycosides (aikacin), second generation fluorquinolones; Response to empirical antibiotic therapy within 72 hours, without modification of empirical antibiotic therapy and without the use of Pentablobin; Response to empirical antibiotic therapy within 72 hours with the use of Pentaglobin within 72 hours of the onset of fever; Response to empirical antibiotic therapy with modification of the antibiotic (without the addition of antifungal), without the use of Pentaglobin; Response to empirical antibiotic therapy with modification of the antibiotic (without the addition of antifungal), with the use of Pentaglobin; Response of antibiotic therapy with empirical addition of antifungal with or without the use of Pentaglobin; Mortality at 30 days; Mortality at 90 days

Design of the study Prospective, observational, non-interventional study to determine the incidence of febrile batteries from MDR germs in febrile oncohaematological patients.

The study is aimed at the centers belonging to the Italian Society of Pediatric Oncology Hematology (IAEOP). Patients will be enrolled prospectively from the date of activation of the center.

Eligible patients will include patients who develop fever after chemotherapy (either after first diagnosis or relapse) or after hemopoietic stem cell transplantation (TCSE) autologhe or allogenic, managed in ordinary hospitalization, subjected to endovenous antibiotic therapy for at least 72 hours for the treatment of the febrile episode. These patients will be the denominator of the study population. Patients who turn out to have positive hemoculture will represent the cases of the study population. A patient may be enrolled several times in the study both as "denominator/control" (hospitalization and example for several febrile episodes) and as a "case" (second episode of febrile batteriemia). In the latter case, the interval between the conclusion of a febrile episode (stable slibration, negative hemoculture) and the subsequent febrile episode must be at least 7 days. The febrile episodes considered will be only those in ordinary hospitalization (minimum 2 nights of hospitalization) while febrile episodes managed exclusively in day-care (Day-Hospital) or with home, oral or endovenous antibiotic therapy are excluded.

Each participating centre must declare at the opening the standard procedure relating to:

1. Study of colonization: yes, no, method of investigation;
2. Standard antibiotic prophylaxis in acute myeloid leukemia (LLA), acute myeloid leukemia (LMA), non-Hodgkin lymphoma (LNH), allogenic TCSE, autologous TCSE;
3. Standard empirical therapy in non-colonized patient (first 48-72 hours);
4. Use of Pentaglobin (yes/no, criteria for use, dose).

In the study patients, hospitalized by febrile episode in endovenous antibiotic therapy, the following information will be collected: sex, age at the time of the febrile episode, age at diagnosis of the basic disease, type of tumor, stage of treatment in hospitalization, type of transplant, presence or not of transplant disease against the host (only for allogenic transplantation), colonization or not, CVC or not, type of CVC, presence or not of urinary catheter, clinical characteristics of the febrile episode, date onset fever-date end fever, date start-date end of antibiotic therapy, date start-date end antifungal therapy, date start-date end therapy with Pentaglobin, result of haemoculture and antibiogram, number of neutrophils, number of lymphocytes, hypotension (in relation to normal values for age, saturation O2, need or not of hospitalization in intensive care , whether or not fluids are used, ventilatory support, renal replacement therapy, , maximum PCR-value (in the first 72 hours), PCT-value (maximum in the first 72 hours), Galactomanane (maximum value during the episode), β-D glucan (maximum value during the episode), survival at 30 and 90 days, final definition of the infectious episode (FUO, ICD, IMD), and possible toxicity related to antibiotic therapy.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent,- onset of fever after chemotherapy or after hemopoietic stem cell transplantation (TCSE),
* endovenous antibiotic therapy for at least 72 hours for the treatment of the febrile episode.
* ordinary hospitalization scheme
* age < 18

Ages: 1 Month to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients with febrile episodes managed during day-care (Day-Hospital) or with home oral or endovenous antibiotic therapy will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-04-22 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of febrile bacteremia due to Gram-negative germs multi-resistant to antibiotics (MDR) | 2020-2023
  The evaluation of the incidence of febrile bacteremia due to MDR Gram-negative germs, i.e. bacteria that present resistance to at least 3 of the 5 classes of main antibiotics (3rd and 4th generation cephalosporins, beta-lactams, aminoglycosides, carbapenems and quinolones).

SECONDARY OUTCOMES:
Incidence of various types of febrile episodes | 2020-2023
  Incidence of various types of febrile episodes: fever of unknown origin (FUO), microbiologically determined infection (MDI) with positive blood culture and without positive blood culture, clinically determined infection (CDI).
  The incidence of the various types of febrile episodes was obtained as the ratio of cases of FUO, IMD with and without bacteremia, fungemia and CDI to total febrile episodes
Bacteremia | 2020-2023
  Incidence of bacteremia due to Gram-negative germs and bacteremia due to Gram-positive germs. The incidence of Gram-negative bacteremia and Gram-positive bacteremia was calculated by the ratio of different events to total IMDs with positive blood culture and total bacteremia.
Fungaemia | 2020-2023
  The incidence of fungemia was calculated as the ratio of fungemia cases to total microbiologically determined infection with positive blood culture.
Risk factors for bacteremia and microbiologically documented infection (MDI) | 2020-2023
  Risk factor analysis for incidence for bacteremia and IMD was performed by logistic regression models
Mortality at 30 days | 30 days
  Evaluate clinical responce and mortality at 30 days. Mortality was derived from the ratio of the number of deaths to the total number of eligible patients.
Mortality at 90 days | 90 days
  Evaluate clinical response and mortality at 90 days. Mortality was derived from the ratio of the number of deaths to the total number of eligible patients.

CONTACTS AND LOCATIONS:
Locations (25):
- Italy (25):
  - Azienda Ospedaliera Universitaria Integrata, Verona, Italia
  - Azienda Ospedali Riuniti Presidio "G. Salesi", Ancona
  - AOU Policlinico, Bari
  - Policlinico Sant'Orsola Malpighi Clinica, Bologna
  - Ospedale Regionale, Bolzano
  - Spedali Civili, Presidio Ospedale Dei Bambini, Brescia
  - Ospedale Pediatrico Microcitemico "Antonio Cao", Azienda Ospedaliera Brotzu, Cagliari
  - AOU Policlinico Vittorio Emanuele, Catania
  - Azienda Ospedaliero Universitaria Sant'Anna, Ferrara
  - Azienda Ospedaliero-Universitaria "Anna Meyer", Florence
  - Istituto G.Gaslini, Genova
  - Fondazione IRCCS Istituto Nazionale Tumori, Milan
  - Azienda Policlinico Di Modena, Modena
  - Fondazione MBBM / AO San Gerardo Clinica, Monza
  - A.O.R.N. Santobono - Pausilipon, Napoli
  - Oncoematologia Pediatrica AOU di Padova, Padua
  - ARNAS Civico Di Cristina E Benfratelli, Palermo
  - Azienda Ospedaliero Universitaria Di Parma, Parma
  - Fondazione IRCCS, Policlinico San Matteo, Pavia
  - A.O.U. "S.M. Della Misericordia", Perugia
  - Ospedale Civile Dello Spirito Santo Dipartimento Di Ematologia, Medicina Trasfusionale E Biotecnologie, Pescara
  - IRCCS Ospedale Pediatrico Bambino Gesù Dip.to di Oncoematologia e Terapia cellulare e Genica, Roma
  - IRCCS Ospedale "Casa Sollievo Della Sofferenza", San Giovanni Rotondo
  - AOU Citta' Della Salute E Della Scienza Di Torino, Torino
  - IRCCS Materno Infantile "Burlo Garofolo", Trieste

IPD SHARING:
Plan to Share IPD: No